CLINICAL TRIAL: NCT00351689
Title: Placebo-controlled Assessment of the Effect of a Food Supplement on Skin Protection After Exposure to UV Radiation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: L'Oreal (Industry)
Collaborators: Société des Produits Nestlé (SPN) (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1030740
Record Dates: First submitted 2006-07-12; First posted 2006-07-13 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Photobiology
Keywords: Probiotic bacteria; cutaneous immune homeostasis; UV radiation; dietary supplement
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: dietary supplement

SUMMARY:
A probiotic bacterial strain was tested in a randomized, double blind , placebo controlled clinical trial with 54 healthy male volunteers. Half the volunteers received the dietary supplement the other half placebo during 6 weeks prior to exposure to solar-simulated UV irradition (2x1,5MED). Blister roofs and skin biopsies were recovered 1, 4 and 10 days after UV exposure from unirradiated and irradiated skin and used for immunohistochemical analysis and mixed epidermal cell lymphocyte reaction

DETAILED DESCRIPTION:
Langerhans cells (LC), the dendritic cells (DC) from epidermis, constitute the first line of immune defense against environmental attacks. Under steady state conditions, LC turnover is very low. The LCs reside in the epidermis in an immature state and can be distinguished from other epidermal cells by their surface expression of HLA-DR, CD1a and langerin. Upon stimulation by inflammatory mediators LCs are activated and acquire CCR7 expression, the chemokine receptor for CCL21 that mediates their migration to lymph nodes. Moreover, activated LCs display a mature phenotype characterized by increased expression of co-stimulatory molecules and acquisition of maturation markers that facilitate their interaction with T-cells and aid in the elicitation of the immune response.

It has long been known that, in addition to being carcinogenic via DNA damage and mutations, solar UV radiation induces local and systemic immune suppression which represents a major risk for skin cancer induction and progression in sun-exposed areas. The process is mostly related to direct LC damage through induction of apoptosis and impairment of antigen-presenting function. Moreover, UV radiation elicits an inflammatory response and subsequent recruitment of immune cells, including CD36+ monocytic cells. These cells colonize the epidermis in the days following UV exposure and are the major source of immunosuppressive cytokines such as IL-10. All these mechanisms ultimately lead to impaired cell-mediated reactions and establishment of immune tolerance.

Nutritional intervention, particularly with dietary antioxidants and vitamins, has been proposed to protect against UV-induced skin damage and to a certain extent skin cancer occurrence. In recent years, there has been an increasing interest for probiotics, defined as live microorganisms which, when consumed in adequate amounts, confer a health benefit upon the host. Particular focus has been on species of lactic acid bacteria including Lactobacilli and Bifidobacteria that are part of the natural human intestinal microbiota. Indeed, it is well documented that the endogenous intestinal microbiota plays a crucial role in immune maturation, gut integrity and defense against pathogens. Recently, it has been shown that some probiotic bacteria possess the ability to modulate the immune system at both the local and systemic levels and thereby improve immune defense mechanisms and/or down-regulate immune disorders such as intestinal inflammations or allergies.

The Probiotic used as the dietary supplement, was isolated from healthy adult microbiota and was shown to have a strong anti-pathogenic activity against a wide range of entero-pathogens. Furthermore, a pre-clinical study demonstrated that it can maintain the epidermal LC density.

Here, we analyzed, in a randomized double blind, placebo controlled, clinical trial, whether this dietary supplement could also modulate the cutaneous immune homeostasis after solar-simulated UV exposure in humans.For this purpose, we analyzed whether this dietary supplement could interfere with LC allostimulatory function and activation/maturation phenotypic status of skin DC, after solar-simulated UV irradiation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject
* Gender: male.
* Age: greater than 20 years and less than 40 years.
* Phototype: II or III.
* Subject having freely given his informed written consent.
* Cooperative subject, aware of the necessity for and duration of the controls, suggesting complete compliance with the protocol set up by Laboratoire DERMSCAN.
* Subject with Social Security coverage.
* A priori, a low fermented milk product consumer (less than 125 g/d) who, during the study, agrees not to eat fermented milk products containing live bacteria (yogurt, cream cheese, fermented dairy products, unpasteurized cheese, etc.).

Exclusion Criteria:

* Subject deprived of freedom by a court or administrative order.
* Minor or major protected by law.
* Subject residing in a health or social care establishment.
* Patient in an emergency setting.
* Subject presenting with skin disease on the test zones.
* Subject presenting with a stable or progressive serious disease (investigator's assessment).
* Immunocompromised subject.
* Subject allergic to one of the constituents of the test products or to xylocaine.
* Subject with a history of allergy to solar or UV radiation.
* Immoderate use of alcohol (more than 2 glasses of wine daily or more than 1 glass of spirits daily).
* Immoderate smoker (more than 6 cigarettes/day).
* Subject exposed to the sun or UV radiation in the last 3 months (facial exposure was authorized with use of a total-block sunscreen and sunglasses).
* Subject with cardiovascular or circulatory disease history.
* Subject with a history of skin cancer, malignant melanoma.
* Subject with a history of intestinal surgery.
* Antibiotic, corticosteroid, non-steroidal anti-inflammatory or immunosuppressant intake.
* Strenuous sports (> 5 hours per week) or naturism.
* Subject having taken a course of mineral supplements or vitamins in the 3 months preceding study initiation.
* Vegetarian or vegan diet.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50
Dates: Start 2004-01; Study Completion 2004-07

PRIMARY OUTCOMES:
Evaluation of food supplement effect on the functions of epidermal cells after UV radiation exposure.

SECONDARY OUTCOMES:
Qualitative analysis (activation and/or maturation status) of cutaneous Langerhans cells and macrophages and analysis of their location and Evaluation of the erythema, pigmentation after UV exposure, Evaluation of safety.

CONTACTS AND LOCATIONS:
Overall Officials: AUDREY GUENICHE, PhD, Study Director — L'Oreal; TIMO BUETLER, PhD, Study Director — Société des Produits Nestlé (SPN)
Locations (1):
- Dermscan, Lyon Villeurbane, France